CLINICAL TRIAL: NCT06004310
Title: Effect of Pulmonary Rehabilitation Among Post-COVID-19 Patients in a Tertiary Care Hospital in Bangladesh: A Quasi-Experimental Study
Brief Title: Effect of Pulmonary Rehabilitation Among Post-COVID-19 Patients in a Tertiary Care Hospital in Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Prof Mohammed Atiqur Rahman, Chairman, Department of Respiratory Medicine, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 683
Record Dates: First submitted 2023-08-17; First posted 2023-08-22 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Pulmonary Pathology
Keywords: Pulmonary rehabilitation,Post-COVID-19 patients,Bangladesh

STUDY DESIGN:
Intervention Model Description: The study will be a quasi-experimental study and carried out at Bangabandhu Sheikh Mujib Medical University. A consecutive sampling method will be used. The participants will engage in a comprehensive 06-weeks outpatient multimodal and multidisciplinary pulmonary rehabilitation program.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post-COVID-19 Patients (Experimental): Post-COVID-19 patients are individuals who have recovered from the acute phase of COVID-19 but continue to experience lingering symptoms and health challenges for weeks or even months after their initial infection. These individuals are often referred to as "long haulers" or "post-acute sequelae of SARS-CoV-2 infection" (PASC) patients. The symptoms experienced by post-COVID-19 patients can vary widely and may include fatigue, shortness of breath, chest pain, joint pain, cognitive difficulties, and more. Medical professionals and researchers are working to better understand and address these conditions, providing supportive care and rehabilitation to help these patients regain their health and well-being.
  Interventions: Behavioral: Pulmonary Rehabilitation

INTERVENTIONS:
Behavioral: Pulmonary Rehabilitation — Participants will be participated a 06 weeks comprehensive outpatient pulmonary rehabilitation which includes endurance training, strength training, patient education, relaxation techniques, psychological support and nutritional counselling.

SUMMARY:
This quasi-experimental study aims to evaluate the efficacy and safety of pulmonary rehabilitation in post-COVID-19 patients and compare differences in primary outcomes before and after pulmonary rehabilitation. Its main aim is to provide an answer to the following question: What are the outcomes of pulmonary rehabilitation in post-COVID-19 patients in a tertiary care facility in Bangladesh? The participants will participate in 06 weeks of comprehensive multimodal and multidisciplinary outpatient pulmonary rehabilitation, including endurance training, strength training, patient education, relaxation techniques, psychological support, and nutritional counseling.

DETAILED DESCRIPTION:
Background: The 2019 novel coronavirus, belonging to the β species of coronaviruses, primarily spreads through respiratory droplets and close contact. Even after recovering from the infection, COVID-19 can lead to various chronic health issues, with impaired lung function, reduced exercise performance, and diminished quality of life being prevalent among a significant proportion of patients. In Bangladesh, post-COVID-19 patients represent a considerable population who have overcome the acute phase of the infection but continue to face numerous social, psychological, and physical challenges. Among these challenges, respiratory complications such as persistent cough, shortness of breath, and decreased lung function are frequently observed in post-COVID-19 patients in Bangladesh. In addition, these individuals often experience fatigue, muscle weakness, and joint pain. These physical symptoms can profoundly impact their daily activities and overall quality of life, necessitating ongoing medical care and rehabilitation.

Purpose: To evaluate the efficacy of pulmonary rehabilitation in post-COVID-19 patients and to compare differences in outcomes between before and after pulmonary rehabilitation Methodology: It will be a hospital-based quasi-experimental study. The investigator will conveniently select adult post-COVID-19 patients whose respiratory symptoms (fatigue, exertional dyspnea, etc.) persist longer than 12 weeks from the onset of their first symptoms from outpatient and inpatient of the Department of Respiratory Medicine, Bangabandhu Sheikh Mujib Medical University. Participants will participate in a 06-weeks (Two sessions per week) comprehensive multimodal and multidisciplinary outpatient pulmonary rehabilitation. In-person interviews will be done for data collection. The total sample size will be 130. Before the study, the research protocol will be approved by the Institutional Review Board (IRB) of Bangabandhu Sheikh Mujib Medical University (BSMMU), Dhaka.

Expected outcome: The study's findings will reveal the benefits of pulmonary rehabilitation among post-COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* Previously RT-PCR positive for SARS-COV-2 and whose respiratory symptoms (fatigue, exertional shortness of breath and cough) persists more than 3 weeks after the onset of their first symptoms attending outpatient and admitted inpatient under the department of Respiratory Medicine, Bangabandhu Sheikh Mujib Medical University, Bangladesh

Exclusion Criteria:

* RT-PCR negative but respiratory symptoms (fatigue, exertional shortness of breath and cough) persists more than 3 weeks after the onset of their first symptoms
* RT-PCR positive but respiratory symptoms (fatigue, exertional shortness of breath and cough) not persists more than 3 weeks after the onset of their first symptoms
* Comorbidities like chronic lung disease, obstructive sleep apnea, coronary heart disease, chronic kidney disease, stroke

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
Distance: Six-minute walking test (6MWT) | After enrollment and after 6 weeks when complete the pulmonary rehabilitation
  The following equipment will be required:
  Stopwatch, Measuring/trundle wheel to measure distance covered, A 30-meter stretch of unimpeded walkway, Two cones to mark the space that needs to be covered, Pulse oximeter for measuring heart rate and SpO2, Borg Breathlessness Scale
Respiratory outcomes: FVC, FEV1, FEV1/FVC ratio, DLCO | After enrollment and after 6 weeks when complete the pulmonary rehabilitation
  FVC (Forced vital capacity) - This is the amount of air exhaled forcefully and quickly after inhaling as much as patient can.
  FEV1 (Forced expiratory volume in 1 second ) - The maximum amount of air that the subject can forcibly expel during the first second following maximal inhalation.
  FEV1/FVC ratio - The ratio of the forced expiratory volume in the first one second to the forced vital capacity of the lungs DLCO (Diffusing lung capacity for carbon monoxide) - The ability of the lungs to transfer gas from inhaled air to the red blood cells in pulmonary capillaries.
Quality of life: Short Form 36 Health Survey Questionnaire (SF-36) | After enrollment and after 6 weeks when complete the pulmonary rehabilitation
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures.
Laboratory investigations: CRP and D-dimer | After enrollment and after 6 weeks when complete the pulmonary rehabilitation
  CRP (C reactive protein) - A c-reactive protein test measures the level of c-reactive protein (CRP) in a sample of patient's blood D-dimer - A D-dimer test looks for D-dimer in blood. D-dimer is a protein fragment (small piece) that's made when a blood clot dissolves in body.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Rahman, MBBS,MD,FCCP, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Shahbag, Bangladesh

IPD SHARING:
Plan to Share IPD: No